CLINICAL TRIAL: NCT05891015
Title: Exploring the Mechanism of Mindfulness Intervention to Alleviate Emotional Distress in Patients With Emotional Disorders
Brief Title: The Mechanism of Mindfulness Intervention to Alleviate Emotional Distress in Patients With Emotional Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Xinghua Liu, Director, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E20230525
Record Dates: First submitted 2023-05-26; First posted 2023-06-06 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Emotional Distress; Emotional Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MIED+TAU group (Experimental): Mindfulness Intervention for Emotional Distress (MIED) program provide standard audio instructions for mindfulness exercises, introduce the nature and law of anxiety, depression and other emotions, the source of anxiety, depression and other emotional distress, and the strategies and methods to alleviate emotional distress. These exercises, knowledge and strategies are based on the latest progress in the field of psychological counseling and treatment, and their application in daily life can help alleviate anxiety, depression and other emotional problems.
  Interventions: Behavioral: Mindfulness Intervention for Emotional Distress(MIED)
- the TAU-only group (No Intervention): treatment as usual (TAU) group consisted of all medicinal and psychological treatments received between baseline and follow-up (about five months). Medicinal treatments included receiving Lorazepam, Olanzapine, Paroxetine Hydrochloride, Sertraline, etc. Psychological treatments included receiving cognitive behavior therapy or psychodynamic therap

INTERVENTIONS:
Behavioral: Mindfulness Intervention for Emotional Distress(MIED) — Mindfulness Intervention for Emotional Distress (MIED) program provide standard audio instructions for mindfulness exercises, introduce the nature and law of anxiety, depression and other emotions, the source of anxiety, depression and other emotional distress, and the strategies and methods to alleviate emotional distress. These exercises, knowledge and strategies are based on the latest progress in the field of psychological counseling and treatment, and their application in daily life can help alleviate anxiety, depression and other emotional problems.
  Arms: MIED+TAU group

SUMMARY:
This study hopes to:

1. explore whether offline and online mindfulness interventions can significantly alleviate individual emotional distress,experiential avoidance and improve cognitive flexibility,distress tolerance level.
2. explore whether cognitive flexibility, distress tolerance and experiential avoidance are the mediators in mindfulness intervention to alleviate emotional distress, and to meet the principles of mechanism.

DETAILED DESCRIPTION:
Cognitive flexibility is a component of executive function, which refers to the ability to transform cognitive models to adapt to changing environmental needs.Empirical avoidance refers to an individual's resistance to experience or attempts to eliminate certain experiences (such as emotions, thoughts, physical sensations, memories, behavioral tendencies, etc.) and attempts to adopt corresponding strategies to change these experiences and the situations in which they are generated. Distress tolerance to negative emotions is considered to be one of the most important cross-diagnostic predictors of emotional distress.

Studies have shown that people with less cognitive flexibility are less effective at using cognitive restructuring techniques to alleviate emotional distress than those with better cognitive flexibility, which seems to predict the level of cognitive flexibility. Cognitive flexibility levels at the three-month follow-up period were significantly negatively correlated with depression levels and suicidal ideation, and higher levels of cognitive flexibility at baseline significantly predicted lower levels of depression and suicidal ideation in military personnel at the three-month follow-up period. Task switching task was used to measure emotional cognitive flexibility, and explored whether individual differences in cognitive flexibility predicted higher levels of trait anxiety and worry within seven weeks. The results showed that emotional cognitive flexibility in the baseline period seemed to predict anxiety and worry levels after seven weeks.

There is a significant positive correlation between mindfulness and cognitive flexibility. One study compared the changes of cognitive flexibility between the mindfulness based cognitive therapy (MBCT) intervention group and the waiting control group in a randomized controlled study of patients with mild to moderate depression. The results showed that the self-reported cognitive flexibility of the MBCT intervention group was significantly higher than that of the waiting control group, and was significantly correlated with the relief of depressive symptoms.

Some reviews suggest that empirical avoidance is one of the mechanisms for the beneficial effects of mindfulness. Some cross-sectional studies suggest that reduced empirical avoidance is an important mediating factor in the mindfulness to psychopathology pathway, a recent cross-sectional study tested the scales of mindfulness, experiential avoidance and anxiety among college students, and the results showed that experiential avoidance could significantly mediate the relationship between trait mindfulness and anxiety, while trait mindfulness could not mediate the relationship between experiential avoidance and anxiety.

Some distress tolerance related variables, such as uncertainty tolerance and experiential avoidance, were found to mediate between mindfulness or mindfulness interventions and emotional distress.

Generally speaking, exploring the mechanism of the effect of mindfulness-based intervention on emotional distress is helpful to strengthen the positive components of the intervention to optimize the therapeutic effect, distinguish the specificity of treatment from the broader non-specific effect, promote the identification of therapeutic regulators and the matching of therapeutic individuals, and provide information for theoretical development and interpretation of results. With the rapid development of online projects and online platforms, online mindfulness courses begin to receive more and more attention, and show a good application prospect. However, there are few studies on online mindfulness courses at present. In order to better understand the effectiveness of online mindfulness courses, more randomized controlled trials need to be done in the future. Therefore, this study will explore the effect of mindfulness intervention on emotional distress and the mechanism of cognitive flexibility, empirical avoidance and distress tolerance based on the basic criterion to judge the mechanism of psychological intervention.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with scores greater than 21 on the Kessler Psychological Distress Scale.
* Subjects have been diagnosed emotional disorders in the past 6 months.

Exclusion Criteria:

* Subjects who could not access the Internet;
* Subjects with insufficient Chinese ability;
* Subjects who have participated in mindfulness based projects for more than 6 weeks before, and / or the current frequency of meditation practice is more than once a week;
* Patients with schizophrenia or psychotic affective disorder, current organic mental disorder, substance abuse disorder and generalized developmental disorder;
* Subjects at risk of suicide.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-06-20 (Estimated); Primary Completion 2023-11-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Weekly changes of Five Facet Mindfulness Questionnaire during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  The Five Facet Mindfulness Questionnaire is a self-reported questionnaire measuring mindfulness levels. Scores range from 39 to 195, with higher scores indicating higher levels of mindfulness.
Weekly changes of Patient Health Questionnaire during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  The Patient Health Questionnaire is a self-reported questionnaire measuring the degree of being troubled by various common physical symptoms. Scores range from 0 to 30.0~4 scores: no physical symptoms; 5~9 scores: mild physical symptoms; 10~14 scores: moderate physical symptoms; 15~30 scores: severe physical symptoms.
Weekly changes of Chinese Perceived Stress Scale during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  The Chinese Perceived Stress Scale is a self-reported questionnaire measuring stress. Scores range from 0 to 56, with higher scores indicating higher levels of stress.
Weekly changes of 10-item Kessler Psychological Distress Scale during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  The 10-item Kessler Psychological Distress Scale is a self-reported questionnaire measuring distress. Scores range from 10 to 50, with higher scores indicating higher levels of distress.
Weekly changes of Overall Anxiety Severity and Impairment Scale during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  The Overall Anxiety Severity and Impairment Scale is a self-reported questionnaire measuring anxiety. Scores range from 0 to 20, with higher scores indicating higher levels of anxiety.
Weekly changes of Overall Depression Severity and Impairment Scale during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  The Overall Depression Severity and Impairment Scale is a self-reported questionnaire measuring depression. Scores range from 0 to 20, with higher scores indicating higher levels of depression.
Weekly changes of Inner Peace Scale during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  The Inner Peace Scale is a self-reported questionnaire measuring peace. Scores range from 0 to 28, with higher scores indicating higher levels of peace.
Weekly changes of Athens Insomnia Scale during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  The Athens Insomnia Scale is a self-reported questionnaire measuring sleepy quality. Scores range from 0 to 24, with lower scores indicating higher levels of sleep quality.
Weekly changes of 16items Chinese Version of the Attentional Control Scale during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  6items Chinese Version of the Attentional Control Scale is a self-reported questionnaire measuring attentional control level.Scores range from 16 to 64, with higher scores indicating higher levels of Attentional Control.
Weekly changes of Cognitive flexibility Inventory during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  Cognitive flexibility Inventory is a self-reported questionnaire measuring Cognitive flexibility level.Scores range from 20 to 100, with higher scores indicating higher levels of Cognitive flexibility.
Weekly changes of Decentralized Questionnaire during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  Decentralized Questionnaire is a self-reported questionnaire measuring decentralization ability. Scores range from 20 to 100, with higher scores indicating higher levels of Decentralized ability.
Weekly changes of Beck Depression Inventory during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  Beck Depression Inventory is a self-reported questionnaire measuring depression level.Scores range from 0 to 63, with higher scores indicating higher levels of depression.
Weekly changes of Beck Anxiety Inventory during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  Beck Anxiety Inventory is a self-reported questionnaire measuring Anxiety level.Scores range from 0 to 63, with higher scores indicating higher levels of Anxiety.
Weekly changes of Ruminative Responses Subscale during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  Ruminative Responses Subscale is a self-reported questionnaire measuring Ruminative Responses level.Scores range from 22 to 88, with higher scores indicating higher levels of Ruminative Responses.
Weekly changes of Emotion Regulation Questionnaire during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  Emotion Regulation Questionnaire is a self-reported questionnaire measuring cognitive reappraisal level.Scores range from 6 to 42, with higher scores indicating higher levels of cognitive reappraisal ability.
Weekly changes of Automatic thoughts questionnaire during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  Automatic thoughts questionnaire is a self-reported questionnaire measuring Automatic thoughts level.Scores range from 30 to 160, with higher scores indicating higher levels of Automatic thoughts.
Weekly changes of Cognitive biases questionnaire during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  Cognitive biases questionnaire is a self-reported questionnaire measuring Cognitive biases level.The score compares the scores of four depression-distortion combinations on a scale of 0 to 23.
Weekly changes of Thought suppression scale during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  Thought suppression scale is used to measure the degree of inhibition of an individual's thinking.Scores range from 15 to 75, with higher scores indicating higher levels of thought suppression.
Weekly changes of Chinese version of the Brief Experiential Avoidance Questionnaire during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  Chinese version of the Brief Experiential Avoidance Questionnaire scale is used to measure Experiential Avoidance.Scores range from 15 to 90, with higher scores indicating higher levels of experiential avoidance.
Weekly changes of Acceptance and Action Questionnaire-II during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  Acceptance and Action Questionnaire-II is used to measure Experiential Avoidance.Scores range from 7 to 49, with higher scores indicating higher levels of experiential avoidance.
Weekly changes of Distress Tolerance Scale during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  Distress Tolerance Scale is used to measure Distress Tolerance.Scores range from 5 to 75, with higher scores indicating higher levels of Distress Tolerance.

SECONDARY OUTCOMES:
Task Switching Task | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  The measurement of cognitive flexibility comes from the task switching paradigm, in which participants are required to classify emotional images according to "emotional task rules" or "non-emotional task rules". In emotional task rules, participants are instructed to classify images according to whether the depicted scene is positive or negative. For non-emotional task rules, participants must indicate whether the number of people in the graph is one or none (≤ 1), or two or more (≥ 2). Even if there is only a part of a person's body, it counts. The image is taken from the International emotional Image system (International Affective Picture System,IAPS). There are 40 pictures in each category: ≤ 1 person + positive, ≥ 2 + positive, ≤ 1 person + negative, ≥ 2 + negative, a total of 160 pictures. Positive and negative images differ in titer ratings, but are balanced in evocative ratings. Another 20 pictures are used for the practice module.
Image rating task | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  The participants were asked to rate their emotional responses to positive, negative and neutral images presented by the computer, and secretly recorded the rated responses
The Paced Auditory Serial Addition Task-Computerized; PASAT-C | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  In this task, participants were presented with a series of numbers and were given the task of adding the last two numbers. They were given points for correct answers and unpleasant vocal feedback for incorrect answers.The task consists of four stages: (1) simple stage, which is the control condition of cognitive and motor function; (2) Latency test stage to determine the level of completion of the addition test; (3) pain induced stage, used to induce emotional pain; (4) Pain tolerance stage, used to measure pain tolerance (i.e. the time before task termination).
Emotional Image Tolerance Task | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  In this task, a series of emotional graphs will be presented on the screen, and the individual needs to first judge whether the picture induces pain. If it does, the duration of the individual's persistence before jumping to the next picture will be taken as the behavioral index of distress tolerance.

CONTACTS AND LOCATIONS:
Overall Officials: Xinghua Liu, Principal Investigator — School of Psychological and Cognitive Sciences, Peking University
Locations (1):
- Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No